CLINICAL TRIAL: NCT03253822
Title: The Effect of a Colorectal Cancer Screening Decision Aid Tailored for People With Lower Educational Attainment in the Central Denmark Region on Colorectal Cancer Knowledge and Colorectal Cancer Screening Attitude and Participation Rate
Brief Title: The Effect of a Colorectal Cancer Screening Decision Aid Tailored to Lower Educational Attainment Citizens
Acronym: LEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Pernille Gabel, M.D. PhD Fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2012-58-006--1-16-02-94-16
Record Dates: First submitted 2017-07-13; First posted 2017-08-18 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Decision Making; Knowledge, Attitudes, Practice
Keywords: Colorectal Neoplasms; Decision Support Techniques; Early Detection of Cancer; Educational Status; Decision Making; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior; Colorectal Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: The LEAD trial is conducted as a two arm, randomised controlled trial nested into a population-based, organized CRC screening programme conducted in the Central Denmark Region. Citizens who are scheduled to be invited for CRC screening within the study period will be randomly allocated into one two study arms. Further, a historic study arm will be included, in order to be able to assess the effect of receiving the baseline questionnaire:
  1. To receive the DA along with the screening reminder and to receive both baseline and follow-up questionnaires (intervention group)
  2. To receive both baseline and follow-up questionnaires (control group)
  3. To receive a questionnaire comprisng scales from both baseline and follow-up questionnaires (historic cohort)
  Regardless of study arm, all citizens receive standard CRC screening information material according to the CRC screening program procedures.
Masking Description: Since baseline questionnaire is filled out before randomizasion, and citizens will know if they receive the DA or not, participants will not be masked.
  No care providers are involved in the screening program in the phases we study (invitation, reminder, and stool sample), hence no masking in this groups.
  The outcomes are assessed via questionnaire data or from registries (Statistics Denmark and the screening IT system), and no masking is necessary in neither investigators nor outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): This group receives a baseline questionnaire before their screening invitation. Respondents are included, and those receiving a screening reminder receive the decision aid.
  At least three months after their screening invitation the included citizens (baseline questionnaire respondents) will receive a follow-up questionnaire.
  Interventions: Other: Decision aid
- Control group (No Intervention): This group receives a baseline questionnaire before their screening invitation. Respondents are included. At least three months after their screening invitation, baseline questionnaire respondents will receive a follow-up questionnaire.
- Historic cohort (No Intervention): A group of people already invited for colorectal cancer screening. This group receives a questionnaire at least three months after their screening invitation. Respondents are included in the study.

INTERVENTIONS:
Other: Decision aid — The DA is an online tool. The web-based design opens up possibilities to feature more advanced functions, e.g. questions for the participant during the process, and a summary of answers at the end. The DA is tailored to lower educational attainment citizens, and is designed to embrace different information needs in the target population, ranging from a desire to receive a clear recommendation and a minimum of information to the desire to receive full information and make a personalized choice.
  Other Names: DA
  Arms: Intervention group

SUMMARY:
The aim of the trial is to test the effect of a web-based decision aid (DA) on colorectal cancer (CRC) knowledge, decisional conflict, participation rate, and informed choice (evaluated based on knowledge, attitudes and actual participation).

The study includes three study arms. Citizens to be recruited are identified from the Danish Civil Registration System based on residence (Central Denmark Region), age (50-74 years old), and month of birth. A random sample of 15,000 citizens born in December (invited for CRC screening through October/November/December 2017) (study arm 1+2) and 5,000 citizens born in October (invited for CRC screening in January/February 2017) (study arm 3) is identified.

Citizens in study arm 1+2 will receive a baseline questionnaire assessing knowledge, attitudes, worry, and health literacy. Non respondents will receive one reminder after two weeks and after four weeks non-respondents will receive a phone call, offering them to fill out the questionnaire via the phone. Baseline questionnaire respondents are included in the study, and will be randomized into two study arms (intervention group and control group).

Citizens in the intervention group will be identified in the screening IT system. Date of screening invitation and screening reminder (citizens who do not return a stool sample within 45 days of the screening invitation) is retrieved. Citizens receiving a screening reminder will receive a link for the DA. Follow-up questionnaire will be sent to all included citizens in study-arm 1+2 three months after the last screening invitation has been sent out. Citizens have six weeks to respond to the questionnaire.

Study arm 3 is a historic cohort. The citizens receive only one questionnaire at the same time as the baseline questionnaires are sent out to the intervention and control groups. The citizens are included if they respond to the questionnaire within six weeks. Questionnaire reminders are sent out at two and four weeks.

Data on screening invitation date, screening reminder date, returning a stool sample and result will be retrieved from the screening IT system for all included citizens (Study arm 1-3). Lastly, data from Statistics Denmark (on socio-demographic and socio-economic factors) will be included.

DETAILED DESCRIPTION:
Study setting The Danish national colorectal cancer (CRC) screening programme was implemented in Denmark in March 2014. All citizens aged 50-74 years are invited to take up CRC screening biennially, however, the first prevalence round is carried out during a four year period (2014-2017). During the this period, citizens are invited according to month of birth, except citizens aged 49 who are invited just before they turn 50 and citizens turning 75 who are invited prior to their 75th birthday, if they were not invited earlier in the program.

Politically and organisationally the CRC screening programme is nationally directed, but the administrative responsibility is placed within the five regions in Denmark. The Department of Public Health Programmes is responsible for the administration of the CRC screening programme in the Central Denmark Region (CDR).

The CDR has 1.3 million citizens (23% of the total population) of which roughly 390 000 citizens are 50-74 years of age. The citizens receive an invitation, containing a screening kit. The screening test (collection of a stool sample) is performed in the citizen's own home. The stool sample is sent to the clinical biochemical department at the hospital. If the citizens do not return a stool sample within 45 days after receiving the invitation, a screening reminder is received. Citizens, who still do not return a stool sample, are automatically referred to the next screening round, and will receive another invitation two years later. Citizens with a negative test are automatically referred to the next screening round. Citizens with a positive test are invited to have a colonoscopy.

Since 2010, national digitisation has occurred in Denmark. Hence, communication to and from Danish authorities occur via digital mail, in the public email platform E-Boks. Danish residents are obliged to order a digital signature (NemID) which is used as a shared log-in for E-boks, public and private online self-services, and online banking. Only disabled citizens (e.g. physical or cognitive impairment) or citizens unable to satisfactorily identify themselves (e.g. migrants with no permanent resident permit) can be exempted from ordering a NemID. As of May 2016 more than 5 million Danish citizens (87.5% of the entire population including children) have access to E-boks. Exemption from digital communication has been granted to 9.8% of Danish Residents aged 45-74 years.

All letters in the CRC screening programme are sent by digital mail, except from invitation letters, which contains a screening kit and are sent by conventional mail. Citizens exempt from digital communication receive conventional letters via a remote printing system.

All invitations and reminders in the screening program are sent out based on lists generated in the administrative CRC screening program IT system, which is linked to the daily updated Danish Civil Registration System, in which all Danish citizens are registered with unique civil registration numbers (CRN) assigned at birth or at immigration. The department of public health programmes is administratively responsible for the screening program IT system.

Study flow The study population will be identified based on data extraction from the Danish Civil Registration System. 10 000 citizens 50-74 years old, living in the Central Denmark Region born in December (invited for CRC screening through October/November/December 2017) and 5 000 citizens 50-74 years old, living in the Central Denmark Region born in October (invited for CRC screening in January/February 2017) are identified.

The 10 000 citizens born in December comprise the population to be randomized (study arm 1 and 2). This group of citizens will receive a baseline questionnaire at the beginning of the study period (before receiving screening invitations). Non-respondents receive a questionnaire reminder after two weeks. After four weeks a telephone call is made offering filling out the questionnaire via telephone. Respondents (at six weeks after receiving the questionnaire) are included in the study and randomized into two groups (intervention and control group). All included citizens are monitored in the screening program IT system, in order to identify date of screening invitation and date of screening reminder. Citizens in study arm one (intervention group) receive a decision aid (DA) on the same day as the screening reminder or the next day. Both groups receive a follow-up questionnaire three months after the date of invitation for the last citizen invited in the study population. Questionnaire reminders are sent out at two and four weeks, and deadline for questionnaire response will be after six weeks.

The 5 000 citizens born in October comprise a historic cohort of citizens invited to CRC screening. This population receives only one questionnaire 3-4 months after they received their screening invitations. In this survey reminders will be sent out at two and four weeks. Respondents (at six weeks) will be included in the study.

All contact with the study participants in this study will occur via digital communication or by postal mail via remote printing system. Hence all questionnaires, survey reminders, and DAs will be sent out first via digital mail. However, it is crucial to reach a high questionnaire participation rate in order to obtain generalizable results. The aim is to reach a survey participation rate of no less than 50% for baseline and 80% for follow-up.

When questionnaire data has been collected, date of screening invitation and screening reminder will be collected from the screening program IT system along with the date of test registration laboratory and the test result.

Questionnaire data and IT system data are both uploaded to Statistics Denmark, where socio-demographic data are appended for the data management and data analysis.

Materials Three different questionnaires will be administered in this trial: The baseline questionnaire, the follow-up questionnaire, and the questionnaire for the historic cohort. The questionnaires comprise five different scales. The worry scale, the knowledge scale, the attitudes scale, the decisional conflict scale, and the health literacy scale, developed by the European Union consortium (HLS-EU-Q16).

The DA is an online tool. The web-based design opens up possibilities to feature more advanced functions, e.g. questions for the participant during the process, and a summary of answers at the end. Further a web-based design has lower running costs, and can be provided as a link via the E-boks platform. The development of the DA took place in five steps: (1) scoping of the DA; (2) formation of the steering group (the research group); (3) Design phase, in which the prototype was developed based on previous research by the research group; (4) Alpha testing, including citizens and experts evaluating design and usability and a peer review by experts and citizens, evaluating content and usability; (5) Beta testing, including citizens, evaluating feasibility, comprehensibility and usability.

The development took place as an iterative process, in which the DA was revise between each step based on the experiences gained from the previous step.

Background data on educational level, family income, occupation, marital status, and ethnicity will be obtained from Statistics Denmark when questionnaire data have been collected.

Statistical methods All statistical analyses are going to be carried out in Stata/SE 14 (STATACorp LP, College Station, Texas, USA), stratifying according to gender. All estimates will be presented with 95% confidence intervals, and all analyses will be carried out on a 5% significance level. Since citizens with lower educational attainment (LEA) are the target group of this study, all citizens with medium or higher educational attainment will be excluded from the statistical analyses.

Pearson's chi-square test will be used to test differences in demographic characteristic distribution between respondents and non-respondents as well as between the study arms in order to test whether the randomisation succeeds.

Differences in distributions of responses to the outcomes (informed choice, yes/no; Adequate knowledge, yes/no; mean level of decisional conflict; mean level of decisional support; mean level of effectiveness of decision made; mean level of worries; and participation, yes/no) in the study arms are being analysed using the independent sample t test for continuous variables and Pearson's chi-square test for categorical variables. Further, the relative risk (RR) will be estimated for all dichotomous outcomes using a 2x2 table with study arm 2 and historic study arm as the reference, respectively.

If randomisation does not succeed in producing groups with similar baseline characteristics, a logistic regression will be completed for categorical outcomes and a linear regression for continuous outcomes in order to estimate an adjusted odds ratio (OR) as a value to be interpreted as a RR.

All analyses will be conducted as intention to treat (ITT) analyses, in which all LEA citizens will remain in the study arms to which they were first assigned.

Power calculations Every month 9 900 citizens are invited to participate in CRC screening in the CDR. On average, 47% of these (4 600) do not return a stool sample within 45 days, and they receive a screening reminder. It is expected that at least 1 200 (26% of the population, according to Statistics Denmark) have LEA. Power calculations (considering a 5% significance level and an 80% statistical power) based on being able to detect expected differences of the outcomes of 22% (proportion making an informed choice), 14% (proportion having a positive attitude towards CRC screening), 16% (proportion participating in CRC screening) and 2.4 (difference in mean score of knowledge) between the groups (as observed in previous studies) indicate that 200 citizens with LEA needs to be included in every group thereby a total of 770 citizens who receive a screening reminder. Analyses are stratified by gender; therefore the study population is doubled to 1 540 participants in every group, so that adequate power is retained to assess the effect of the DA in both genders.

With an expected participation rate of 58% for baseline questionnaire (study arm 1+2) and an expected participation rate of 80% in the follow-up questionnaire in study arms 1 and 2, 10 000 citizens who will be invited for screening (5 000 in each study arm and hence an allocation ratio of 1:1) are included. In the historic study arm a 50% participation rate is expected (two written reminders, no telephone calls), hence we 5 000 citizens, who will be invited for screening, are included.

ELIGIBILITY:
Inclusion Criteria:

* Random sample of citizens 50-74 years of age.
* Resident in the Central Denmark Region at time of data extraction (August 2017)
* Month of birth: December or October

Exclusion Criteria:

* Non-respondents to baseline questionnaire (study arm 1+2) or questionnaire (study arm 3)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15030 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
CRC and CRC screening knowledge | Assessed before screening invitation (study arm 1+2) and at least three months after screening invitation (study arm 1+2+3)
  Assessed using questionnaire. Six items yielding a scale score between 0 and 100 %. Continous variable.
CRC screening attitude | Assessed before screening invitation (study arm 1+2) and at least three months after screening invitation (study arm 1+2+3)
  Assessed using questionnaire. Four items. Scores between 7 and 28. Continuous variable.
CRC screening participation | Obtained at least three months after screening invitation.
  Binary outcome (yes/no), retrieved from screening IT system.

SECONDARY OUTCOMES:
CRC worry | Assessed before screening invitation (study arm 1+2) and at least three months after screening invitation (study arm 1+2+3)
  Assessed in questionnaire. Three items. Individually scored.
Decisional conflict | Assessed at least three months after invitation (study arm 1+2+3)
  Decisional conflict scale. Questionnaire. 16 items. score 0-100 points.
Health literacy | Assessed before screening invitation (study arm 1+2) or at least three months after screening invitation (study arm 3)
  HLS-EU-Q16 scale. Questionnaire. 16 items. Score 0-16.
Educational level | Up to 12 months before screening invitation
  Socio-demographic outcome, Statistics Denmark. LEA (≤10 years of education) and medium or high educational attainment (>10 years of education)
Family income | Up to 12 months before screening invitation
  Socio-demographic outcome, Statistics Denmark.The categories will be lower tertile, middle tertile, and upper tertile.
Occupation | Up to 12 months before screening invitation
  Socio-demographic outcome, Statistics Denmark. Employed, Self-employed chief executive, Unemployed/receiving benefits, Retired, Social welfare recipients, and Others.
Marital status | Up to 12 months before screening invitation
  Socio-demographic outcome, Statistics Denmark. Married/cohabitant or single/widow
Ethnicity | Up to 12 months before screening invitation
  Socio-demographic outcome, Statistics Denmark. Danish, Immigrant (Western origin), and Immigrant (non-western origin)

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Gabel, MD PhD Fel., Principal Investigator — Department of Public Health Programmes, Randers Regional Hospital, Central Denmark Region, Denmark
Locations (1):
- Department of Public Health Programmes, Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No
No individual patient data are to be shared with other researchers.